CLINICAL TRIAL: NCT01966432
Title: Screening, Brief Intervention, and Referral to Treatment in Primary Care (SBIRT-PC): An add-on Project to "Duke University Southeastern Diabetes Initiative"
Brief Title: Screening, Brief Intervention, and Referral to Treatment in Primary Care
Acronym: SBIRT-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00043463_1; 2U10DA013727 (NIH); CTN-0057 OT (Other Grant/Funding Number: National Institute on Drug Abuse); 3UG1DA040317 (NIH)
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2; Substance-related Disorders
Keywords: Substance abuse; Alcohol use; Tobacco use; Brief intervention; Referral to treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Substance-Related Disorders; Alcohol Drinking; Tobacco Use | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: This is a single group, non-randomized, pilot study that explores the feasibility of applying SBIRT to adult with high-risk diabetes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBIRT (Other): This is a single arm, non-randomized study. However, based on participants' substance use status, participants will be categorized into three groups:
  1. Screening group. Patients who screen for no use of cigarettes, alcohol, or other drugs. Patients are re-screened at followup visits.
  2. Screening, Brief Intervention group. Patients who screen positive for cigarette, alcohol, or other drug use.
  3. Screening, Brief Intervention, and Referral to Treatment group. Patients who screen positive for use and have a positive AUDIT-C and/or positive DAST-10 assessment for problematic alcohol or drug use.
  Interventions: Behavioral: Referral to Treatment; Behavioral: Brief Intervention

INTERVENTIONS:
Behavioral: Referral to Treatment — Patients receive a referral to treatment for substance abuse, with up to 2 follow-up phone calls. Patients are re-screened at followup visits.
Behavioral: Brief Intervention — Patients receive a brief intervention aimed at reducing substance use, and are re-screened at followup visits.

SUMMARY:
This add-on study of providing tobacco, alcohol and other drug screening, brief intervention and referral for treatment to a primary care high risk diabetic population leverages the existing research resources of a funded parent project "Duke University CMS Innovation Award Southeastern Diabetes initiative (PI: Robert M. Califf, MD)" to explore the feasibility of implementing Screening for substance use, Brief Intervention, and Referral to Treatment services in Primary Care (SBIRT-PC) and to examine the effects of substance use status on diabetes health care outcomes. This pilot study also examines the feasibility of the CTN's common data element algorithms of SBIRT for illicit and nonmedical drug use in the primary care setting.

DETAILED DESCRIPTION:
Duke University Translational Medicine Institute has received funds from the Bristol-Myers Squibb Foundation and the Centers for Medicare and Medicaid Services (2012-2016) to augment existing standard of care for patients with diabetes in community-based medical settings in order to achieve goals of better health, better health care, and reduced costs ("Duke University CMS Innovation Award Southeastern Diabetes initiative"; Principal Investigator, Robert M. Califf, MD). Its goals are to (1) improve population-level diabetes management, health outcomes, and quality of life for diagnosed and undiagnosed adults living with type 2 diabetes, (2) reduce disparities in diabetes management, health outcomes and quality of life for adults living with type 2 diabetes, and (3) reduce healthcare costs associated with type 2 diabetes. This already funded diabetes care project provides a cost-effective platform for conducting an add-on project to examine the feasibility of the CTN's clinical decision support algorithms for SBIRT in primary care settings, as the study team can leverage existing organizational and research infrastructure to facilitate the completion of the study. The add-on study is supported by strong rationale, including the fact that primary care settings serve as common points of contact for adults and provide many opportunities to detect drug misuse and to intervene early in low or mild severity (better outcomes), which in turn may reduce substance use, increase awareness and drug-medication interactions, enhance patient medication adherence, and decrease high inpatient costs and repeat emergency department visits.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Diagnosis of Type 2 diabetes
* Reside in Durham County, NC, or the neighboring areas and receive the majority of their healthcare in the county
* Referral from the primary care clinician or patient's medical home if one has been designated
* Have capacity to make decisions

Exclusion Criteria:

* Lack capacity to make decisions and do not have a surrogate with authority to make health care decisions.
* Have a terminal illness with a life expectancy of 6 months or less
* Diagnosis of Type 1 diabetes or gestational diabetes
* Currently pregnant
* Unable to comply with study requirement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzy Wu, RN, ScD, Principal Investigator — Duke University
Locations (1):
- Durham County Department of Public Health, Durham, North Carolina, United States

REFERENCES:
- [Background] Wu LT, Brady KT, Spratt SE, Dunham AA, Heidenfelder B, Batch BC, Lindblad R, VanVeldhuisen P, Rusincovitch SA, Killeen TK, Ghitza UE. Using electronic health record data for substance use Screening, Brief Intervention, and Referral to Treatment among adults with type 2 diabetes: Design of a National Drug Abuse Treatment Clinical Trials Network study. Contemp Clin Trials. 2016 Jan;46:30-38. doi: 10.1016/j.cct.2015.11.009. Epub 2015 Nov 10. PMID 26563446
- [Result] Wu LT, Ghitza UE, Batch BC, Pencina MJ, Rojas LF, Goldstein BA, Schibler T, Dunham AA, Rusincovitch S, Brady KT. Substance use and mental diagnoses among adults with and without type 2 diabetes: Results from electronic health records data. Drug Alcohol Depend. 2015 Nov 1;156:162-169. doi: 10.1016/j.drugalcdep.2015.09.003. Epub 2015 Sep 12. PMID 26392231
- [Result] Wu LT, Ghitza UE, Zhu H, Spratt S, Swartz M, Mannelli P. Substance use disorders and medical comorbidities among high-need, high-risk patients with diabetes. Drug Alcohol Depend. 2018 May 1;186:86-93. doi: 10.1016/j.drugalcdep.2018.01.008. Epub 2018 Mar 3. PMID 29554592

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Based on the results of the baseline substance use screen for the parent Southeastern Diabetes Initiative (SEDI) study at the Durham site, participants were categorized into three groups: Minimal-risk Screen (S) Group; At-risk Screen & Brief Intervention (SBI) Group; and, High-risk Screen, Brief Intervention, & Referral to Treatment (SBIRT) Group.
Pre-assignment Details: The clinical team consented 134 adults (84% of the eligible patients) for the SBIRT study. Of the 134 adults consented (enrolled), 36 are not accounted for in the results section (do not have baseline data).
Groups:
- SBIRT Group: Screening, Brief Intervention, and Referral to Treatment group. Patients who screen positive for use and have a positive AUDIT-C and/or positive DAST-10 assessment for problematic alcohol or drug use.
  Referral to Treatment: Patients receive a referral to treatment for substance abuse, with up to 2 follow-up phone calls. Patients are re-screened at followup visits.
  Brief Intervention: Patients receive a brief intervention aimed at reducing substance use, and are re-screened at followup visits.
- SBI Group: Screening and Brief Intervention group. Patients who screen positive for cigarette, alcohol, or other drug use.
  Brief Intervention: Patients receive a brief intervention aimed at reducing substance use, and are re-screened at followup visits.
- S Group: Screening only group. Patients who screen for no use of cigarettes, alcohol, or other drugs. Patients are re-screened at followup visits.
Period: Overall Study
Arm/Group | SBIRT Group | SBI Group | S Group
Started | 10 | 34 | 54
Completed | 5 | 21 | 28
Not Completed | 5 | 13 | 26
Not completed — Lost to Follow-up | 3 | 2 | 5
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Subject Incarcerated | 0 | 0 | 1
Not completed — SBIRT program ended | 1 | 8 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBIRT Group | SBI Group | S Group | Total
Number analyzed (Participants) | 10 | 34 | 54 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 33 | 37 | 80
  >=65 years | 0 | 1 | 17 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (5.8) | 51 (9.1) | 60 (12.0) | 56 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 33 | 54
  Male | 3 | 20 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 9 | 31 | 53 | 93
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 28 | 44 | 80
  White | 1 | 4 | 5 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 34 | 54 | 98

OUTCOME MEASURES:

1. Primary Outcome: Drug Use Status and Frequency
Description: Results of DAST-10 survey to determine use of illicit or nonmedical drugs.The Drug Abuse Screening Test (DAST-10) is a 10-item brief screening tool that assesses drug use, not including alcohol or tobacco use, in the past 12 months. Each question requires a yes or no response, and the tool can be completed in less than 8 minutes. DAST-10 scores on a 10-point scale. A score of 0 indicates no problems and 10 indicates a severe level of problems are associated with drug abuse.
Time Frame: Baseline, Six Month Follow-up
Population: All subjects who completed the assessments were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SBIRT Group | SBI Group | S Group
Number analyzed (Participants) | 10 | 34 | 54
units on a scale
  Baseline | 2.00 [0.57 to 3.43] | 0.03 [0.00 to 0.09] | 0.02 [0.00 to 0.06]
  Followup: number analyzed (Participants) | 5 | 18 | 39
  Followup | 0.60 [0.00 to 1.71] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

2. Primary Outcome: Cigarette Smoking Status and Nicotine Dependence
Description: Results from Fagerstrom Test for Nicotine Dependence. The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
Time Frame: Baseline, Six Month Follow-up
Population: All subjects who completed the assessments were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SBIRT Group | SBI Group | S Group
Number analyzed (Participants) | 10 | 34 | 54
units on a scale
  Baseline | 1.50 [0.02 to 2.98] | 2.91 [2.01 to 3.81] | 0.00 [0.00 to 0.00]
  Follow-up: number analyzed (Participants) | 5 | 18 | 39
  Follow-up | 1.60 [0.00 to 4.84] | 2.78 [1.71 to 3.85] | 0.00 [0.00 to 0.00]

3. Primary Outcome: Alcohol Use Status
Description: Results of AUDIT-C survey. The AUDIT-C is a 3-item alcohol screen that can help identify people who are hazardous drinkers or have active alcohol use disorders. AUDIT-C is scored on a scale of 0-12. The higher the score, the more likely it is that the person's drinking is affecting his/her safety
Time Frame: Baseline, Six Month Follow-up
Population: All subjects who completed the assessments were included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SBIRT Group | SBI Group | S Group
Number analyzed (Participants) | 10 | 34 | 54
units on a scale
  Baseline | 1.60 [0.00 to 4.06] | 0.76 [0.37 to 1.16] | 0.00 [0.00 to 0.00]
  Follow-up: number analyzed (Participants) | 5 | 18 | 39
  Follow-up | 0.00 [0.00 to 0.00] | 0.44 [0.00 to 0.90] | 0.00 [0.00 to 0.00]

4. Primary Outcome: Percentage of Participants Who Reported Substance Use at 6 Month
Description: For SBI and SBIRT groups: Proportion of baseline substance users (SBI, SBIRT) who continue substance use during the study (self reported) For S group: Proportion of baseline non-users (S) who report substance use during follow-up visit
Time Frame: Baseline, Six Month Follow-up
Population: All subjects who completed the assessments were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SBI Group: Screening, Brief Intervention group. Patients who screen positive for cigarette, alcohol, or other drug use.
  Brief Intervention: Patients receive a brief intervention aimed at reducing substance use, and are re-screened at followup visits.
- S Group: Screening group. Patients who screen for no use of cigarettes, alcohol, or other drugs. Patients are re-screened at followup visits.
Arm/Group | SBIRT Group | SBI Group | S Group
Number analyzed (Participants) | 10 | 34 | 54
percentage of participants
  Baseline | 30.0 [10.8 to 60.3] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Followup: number analyzed (Participants) | 5 | 18 | 39
  Followup | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

5. Primary Outcome: Treatment for Drug Use or Alcohol
Description: Percentage of patients who received substance abuse or alcohol treatment (self reported)
Time Frame: Baseline, Six Month Follow-up
Population: All subjects who completed the assessments were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SBIRT Group | SBI Group | S Group
Number analyzed (Participants) | 10 | 34 | 54
percentage of participants
  Baseline | 20.0 [5.7 to 51.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Followup: number analyzed (Participants) | 5 | 18 | 39
  Followup | 20.0 [3.6 to 62.4] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: Adverse Event data collected at baseline interview.
Arm/Group | SBIRT Group | SBI Group | S Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/34 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/34 | 0/54
Other Adverse Events (participants affected / at risk) | 0/10 | 0/34 | 0/54

LIMITATIONS AND CAVEATS:
This pilot study is not randomized, and it is not designed for hypothesis testing. Any conclusions arising from these data must be regarded as exploratory and preliminary, and need to be validated by independent data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No